CLINICAL TRIAL: NCT00712842
Title: Neurovascular Coupling in Patients With Early Stage Diabetes Retinopathy
Status: Completed | Type: Observational
Sponsor: Gerhard Garhofer (Other)
Responsible Party: Sponsor-Investigator, Gerhard Garhofer, MD, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: OPHT-221203
Record Dates: First submitted 2008-07-07; First posted 2008-07-10 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetes; ocular blood flow
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients with non or mild non-proliferative diabetic retinopathy
  Interventions: Other: Ocular blood flow measurements
- 2: Healthy control subjects
  Interventions: Other: Ocular blood flow measurements

INTERVENTIONS:
Other: Ocular blood flow measurements — non-invasive haemodynamic measurements of retinal vessel diameters and laser Doppler velocimetry

SUMMARY:
A variety of studies demonstrate that ocular blood flow is altered in diabetes and retinal perfusion abnormalities have been proposed to contribute to the pathogenesis of diabetic retinopathy.

Various animal and human studies have demonstrated that retinal and optic nerve blood flow increase in response to diffuse luminance flicker. Based on studies with ERG, this effect has been attributed to augmented activity in the retinal ganglion cells and associated axons indicating a coupling mechanism between neuronal activity and retinal blood flow. Whereas a variety of studies describe the effects of flickering light on retinal and optic nerve head blood flow, the knowledge about this coupling in the diabetic retina is sparse.

In view of the fact that neural activity and blood flow are strongly coupled in the human retina, one could hypothesize that neurodegenerative changes in the retina could contribute to the vascular dysregulation and in turn lead to changes of ocular perfusion. The investigators set out to investigate whether the coupling of neural activity and blood flow is impaired in patients with early stage diabetic retinopathy compared to those in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 20 and 50 years
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Inclusion criteria of patients are insulin dependent diabetes mellitus (IDDM) with non or mild non-proliferative retinopathy. Patients with no signs of diabetic retinopathy (level 1) or patients with one or more microaneurysms (level 2) will be included. Duration of Diabetes is between 5 and 20 years
* Men and women will be included in equal parts. A pregnancy test will be performed at screening
* Ametropia of less than 3 diopters and anisometropia of less than 1 diopter

Exclusion Criteria:

* Non insulin dependent diabetes
* Maturity onset diabetes of the young (MODY diabetes)
* Any sign of non diabetes induced vascular pathologies, systemic hypertension (defined as systolic blood pressure > 150 mm Hg and diastolic blood pressure > 90 mm Hg.)
* Presence of intraocular pathology other than diabetic retinopathy
* History or family history of epilepsy
* Pregnancy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 50 Patients with Diabetes Type 1 50 Healthy Control Subjects
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-01; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | 90 minutes
Retinal arterial and venous diameter | 90 minutes
Retinal blood velocity | 90 minutes
Pattern ERG | measured once on the study day

SECONDARY OUTCOMES:
Mean arterial pressure | 90 minutes
Blood glucose | measured once on the study day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Lasta M, Pemp B, Schmidl D, Boltz A, Kaya S, Palkovits S, Werkmeister R, Howorka K, Popa-Cherecheanu A, Garhofer G, Schmetterer L. Neurovascular dysfunction precedes neural dysfunction in the retina of patients with type 1 diabetes. Invest Ophthalmol Vis Sci. 2013 Jan 30;54(1):842-7. doi: 10.1167/iovs.12-10873. PMID 23307962